CLINICAL TRIAL: NCT02989896
Title: Evaluation of Perfusion Index in the Success of Peripheral Nerve Block in Advanced Age Patients
Brief Title: Perfusion Index in the Success of Peripheral Nerve Block
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Erzincan University (Other)
Responsible Party: Principal Investigator, ILKE KUPELI, assist. prof., Erzincan University
Other Study IDs: ERZINCAN UNIVERSITY 5
Record Dates: First submitted 2016-12-04; First posted 2016-12-12 (Estimated); Last update posted 2016-12-12 (Estimated); Status verified 2016-12

CONDITIONS: Perfusion Index; Peripheral Nerve Block Success
Keywords: Perfusion index; Peripheral nerve block success; older age
MeSH Terms: interventions — Perfusion Index

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: perfusion index

SUMMARY:
After a successful peripheral nerve block, blockade of sympathetic nerve fibers results in local vasodilatation, increased local blood flow, and increased skin temperature.Increased permeability index; Can be used as a reliable tool for evaluating block activity.

ELIGIBILITY:
Inclusion Criteria:

* Over 65 years old
* ASA I-III

Exclusion Criteria:

* Patients under 65 years old
* Patients contraindicated in regional anesthesia
* Patients with local anesthetic allergy
* Patients with injection site infection
* Patients who do not accept the procedure

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Elective orthopedic lower extremity surgery patients
Sampling Method: Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2016-12; Primary Completion 2017-08 (Estimated); Study Completion 2017-09 (Estimated)

PRIMARY OUTCOMES:
patient's perfusion index | nine month

REFERENCES:
- [Background] Curatolo M, Petersen-Felix S, Arendt-Nielsen L. Sensory assessment of regional analgesia in humans: a review of methods and applications. Anesthesiology. 2000 Dec;93(6):1517-30. doi: 10.1097/00000542-200012000-00025. No abstract available. PMID 11149448
- [Background] Pearson AC, Gudipati CV, Labovitz AJ. Effects of aging on left ventricular structure and function. Am Heart J. 1991 Mar;121(3 Pt 1):871-5. doi: 10.1016/0002-8703(91)90201-r. PMID 1825740
- [Background] Lima AP, Beelen P, Bakker J. Use of a peripheral perfusion index derived from the pulse oximetry signal as a noninvasive indicator of perfusion. Crit Care Med. 2002 Jun;30(6):1210-3. doi: 10.1097/00003246-200206000-00006. PMID 12072670
- [Background] Kus A, Gurkan Y, Gormus SK, Solak M, Toker K. Usefulness of perfusion index to detect the effect of brachial plexus block. J Clin Monit Comput. 2013 Jun;27(3):325-8. doi: 10.1007/s10877-013-9439-4. Epub 2013 Feb 10. PMID 23397432
- [Background] Galvin EM, Niehof S, Verbrugge SJ, Maissan I, Jahn A, Klein J, van Bommel J. Peripheral flow index is a reliable and early indicator of regional block success. Anesth Analg. 2006 Jul;103(1):239-43, table of contents. doi: 10.1213/01.ane.0000220947.02689.9f. PMID 16790660
- [Background] Sebastiani A, Philippi L, Boehme S, Closhen D, Schmidtmann I, Scherhag A, Markstaller K, Engelhard K, Pestel G. Perfusion index and plethysmographic variability index in patients with interscalene nerve catheters. Can J Anaesth. 2012 Dec;59(12):1095-101. doi: 10.1007/s12630-012-9796-3. Epub 2012 Oct 2. PMID 23055034
- [Background] Goldman JM, Petterson MT, Kopotic RJ, Barker SJ. Masimo signal extraction pulse oximetry. J Clin Monit Comput. 2000;16(7):475-83. doi: 10.1023/a:1011493521730. PMID 12580205